CLINICAL TRIAL: NCT07368933
Title: ADVANCEd NanoTherapies SirPlux Duo™ Dual API-Coated PTCA Balloon Catheter to Treat Coronary In-stent Restenosis (ISR) and de Novo Lesions
Brief Title: Advanced NanoTherapies Dual-API DCB to Treat De-Novo and ISR Lesions in Patients With Symptomatic Coronary Artery Disease
Acronym: ADVANCE-DUO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced NanoTherapies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANT-00001
Record Dates: First submitted 2026-01-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Angina (Stable); CAD - Coronary Artery Disease; Unstable Angina; NSTEMI - Non-ST Segment Elevation MI
Keywords: DCB; Drug Coated Balloon; Coronary Artery Disease
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease; Angina, Unstable; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- SirPlux Duo™ Dual API-Coated PTCA Balloon Catheter (Experimental): Subject who meet the inclusion criteria and agree to participate in the study will be enrolled and undergo a planned percutaneous coronary intervention with SirPlux DUO PTCA
  Interventions: Device: SirPlux Duo™ Dual API-Coated PTCA Balloon Catheter

INTERVENTIONS:
Device: SirPlux Duo™ Dual API-Coated PTCA Balloon Catheter — SirPlux Duo PTCA is a Drug-Coated Balloon to treat de novo and In-Stent Restenosis lesions in patients with symptomatic stable angina, unstable angina or NSTEMI

SUMMARY:
The study objectives are:

1. To evaluate the safety and performance of the SirPlux Duo PTCA to treat coronary ISR lesions 2.00-4.00 mm (inclusive) in diameter in patients with symptomatic coronary artery disease.
2. To evaluate the safety and performance of the SirPlux Duo PTCA to treat coronary de novo lesions <3.00 mm in diameter in patients with symptomatic coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years or minimum legal age as required by local regulations.
2. Documented stable or unstable angina, positive functional test, or non -ST elevation myocardial infarction which, in the judgment of the operator, is attributable to disease in coronary vessel or in-stent restenosis, and the patient is deemed an appropriate candidate for PCI in accordance with the applicable guidelines on percutaneous coronary intervention.

   Note: participants with NSTEMI must have enzymes that are trending down or are within normal limits prior to enrollment.
3. Life expectancy >1 year in the Investigator's opinion.
4. Participant is willing and able to cooperate with study procedures and follow-up evaluations.
5. Treatment of only one target lesion required

   1. Tandem lesions treated by a single DCB will be considered one target lesion.
   2. Up to one de novo lesion in a separate vessel may be treated per standard of care at the procedure. Non-target lesions must be successfully treated under the same criteria of the target lesion, before treating the target lesion.
6. Target lesion must be ≤36 mm in length.
7. Target lesion must have a stenosis ≥ 50% and < 100%.
8. Target lesion must have a visually estimated reference vessel diameter of:

   1. ISR lesions: 2.0 to 4.0 mm in diameter (inclusive)
   2. de novo lesions: 2.0 to <3.0 mm in diameter
9. ISR lesions only: target lesion must be within a previous BMS or DES that does not extend >5.0 mm beyond the proximal or distal edge.

Exclusion Criteria:

1. Participant is pregnant, or breastfeeding. Note: Participant of childbearing potential must have a negative pregnancy test within 7 days before procedure.
2. Known hypersensitivity or contraindication to antiplatelet medications (e.g., aspirin; heparin; prasugrel); or a sensitivity to contrast media which cannot be adequately pre-medicated.
3. History of an allergic reaction or significant sensitivity to paclitaxel, sirolimus, or any other analogue or derivative.
4. Platelet count < 100,000 cells/mm³ (i.e., 100 x 109 /L) or > 700,000 cells/mm³ (i.e., 700 x 10 9 /L), or a white blood cell (WBC) count < 3,000 cells/mm³ within 7 days prior to procedure.
5. Renal insufficiency (Serum creatinine level > 2.5 mg/dl (i.e., 221 μmol/L) within 7 days prior to procedure) or failure (dialysis dependent).
6. Evidence of an acute MI within 72 hours of the procedure Note: participants with NSTEMI are allowed, provided enzymes are trending down or are within normal limits prior to enrollment.
7. Previous PCI of the target vessel within 6 months prior to procedure.
8. History of a stroke or transient ischemic attack (TIA) within the prior 3 months to procedure (any prior stroke or TIA, if prasugrel is used).
9. Planned PCI of any vessel within 30 days post-procedure and/or planned PCI of the target vessel within 12 months post-procedure.
10. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months to procedure.
11. History of bleeding diathesis or coagulopathy or will refuse blood transfusions.
12. Documented left ventricular ejection fraction (LVEF) <30% at the most recent evaluation, within the prior 3 months to procedure.
13. Planned surgery that would cause interruption in recommended DAPT duration per current guidelines.
14. Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; or requires additional coronary angiography, IVUS, or other coronary artery imaging procedures.
15. The following criteria related to previous treatments applies based on the type of lesion treated. The participant is excluded in the following circumstances:

    1. ISR lesions: If single-layer ISR, any previous treatment of the target vessel for restenosis. If double- layer ISR, any treatment of the double-layer ISR.
    2. de novo lesions: any previous treatment of the target lesion.
16. Planned PCI of three vessel disease during procedure.
17. Planned treatment of more than one target vessel. Tandem lesions that can be treated by a single DCB are permissible.
18. Target lesion requires treatment with atherectomy, laser, or thrombectomy procedure.
19. Target vessel has other lesions with greater than 50% diameter stenosis based on visual estimate.
20. Target vessel has evidence of thrombus.
21. Target vessel is excessively tortuous, defined as more than one bend >90° to reach target lesion.
22. Target lesion has any of following characteristics:

    1. Lesion location is unprotected in left main coronary artery, internal mammary artery, aorto-ostial, bypass grafts, ostial lesions or within 5 mm of the origin of the left anterior descending or left circumflex.
    2. Involves a side branch >2.0 mm in diameter.
    3. Is severely calcified.
23. The following criteria based on number and type of lesions:

    1. ISR and de novo lesions: target lesion is in the same vessel with a de novo lesion requiring treatment.
    2. ISR lesions: planned treatment of a ≥3 layer ISR lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure rate (TLF) | 12 Months
  Target lesion failure rate (TLF) at 12 months post-procedure

SECONDARY OUTCOMES:
Performance - Device Sucess | Peri-procedural
  Device Success: Defined as successful delivery, balloon inflation, deflation, and retrieval of the intact study device.
Performance - Lesion Success | Peri-procedural
  Defined as achievement of ≤30% residual stenosis (by visual estimate) of the target lesion upon SirPlux Duo PTCA treatment
Performance - Procedural Success | Peri-Procedural through 7 days post-Procedure
  Defined as device and lesion success, and absence of procedural complications following study device inflation (i.e., absence of significant vessel dissection [Grade C or higher] or loss of TIMI 3 flow) through 7 days post-procedure
Late Lumen Loss | 6 months post procedure
  Late Lumen Loss based on QCA
Safety | 24 months post procedure
  1. All Death
  2. Cardiac death
  3. All myocardial infarction (MI), including target vessel myocardial infarction (TVMI)
  4. Ischemia driven target lesion revascularization (TLR) defined as revascularization at the target lesion associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis ≥ 50% by QCA.
  5. Clinically driven target lesion revascularization (cd-TLR) defined as revascularization at the target lesion associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis ≥ 50% by QCA, or revascularization of a target lesion with diameter stenosis ≥ 70% by QCA without either angina or a positive functional study.
  6. Ischemia driven target vessel revascularization (TVR) defined as revascularization at the target vessel associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis ≥ 50% by QCA.
Safety | 24 Months post-procedure
  g. Clinically driven target vessel revascularization (cd-TVR) defined as revascularization at the target vessel associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis ≥ 50% by QCA, or revascularization of a target lesion with diameter stenosis ≥ 70% by QCA without either angina or a positive functional study h. Major adverse cardiac event (MACE) defined as composite of death, MI, or repeat TLR i. Target lesion failure (TLF) defined as composite of cardiac death, TVMI, or TLR j. Target vessel failure (TVF) defined as composite of cardiac death, TVMI, or TVR k. Target lesion thrombosis (TLT) (definite or probable) according to Academic Research Consortium (ARC) definition

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No